CLINICAL TRIAL: NCT00406861
Title: Montelukast as an Alternative or Supplementary Treatment in ENL Reaction in Leprosy
Brief Title: Montelukast in ENL Reaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Leprosy Mission Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMRCERC2004-2007627
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Erythema Nodosum Leprosum; Leprosy
Keywords: reaction; ENL; leprosy
MeSH Terms: conditions — Leprosy | interventions — montelukast

INTERVENTIONS:
Drug: montelukast in treatment of ENL reaction

SUMMARY:
Objective of the trial is to assess the safety and efficacy of Montelukast in treatment of Erythema Nodosum leprosum (ENL) reaction in multibacillary leprosy patients either in combination with prednisolone or alone.

Hypothesis is that montelukast will reduce the severity of ENL reaction in Multibacillary leprosy patients without causing an unacceptably high incidence of adverse effects.

Design is a multicentre hospital-based single-blind prospective trial for leprosy patients with ENL reaction. prior written consent will be taken from the patients who will undergo the trial.

Endpoints are decrease in severity of ENL and absence of new nerve function impairment

DETAILED DESCRIPTION:
Leprosy is still a common medical problem in many countries including Bangladesh, and currently there are at least 3500 leprosy patients in this country at risk of ENL reaction, which is a distressing complication of Multibacillary (MB) leprosy liable to result in permanent disability if not well treated. The drug of choice is either prednisolone ( which often causes adverse effects especially with prolonged use) or thalidomide which is not available in Bangladesh.Clofazimine in high doses is recommended as an alternative but supplies are difficult to obtain. Hence the need for an alternative drug which could be used as a steroid sparing agent or an alternative to steroids in ENL reaction. Montelukast is a leukotriene inhibitor already available on the open market in this country as an immunomodulator, and a small clinical trial with zafirlukast ( very similar drug) suggested that drugs in this group may be effective for ENL.

This is a phase two trial to assess the safety and efficacy of montelukast as an alternative or supplementarry treatment for ENL reaction.

Eligible patients presenting to one of the participating hospitals with ENL reaction will be randomly allocated to one of three groups to receive prednisolone only or prednisolone plus montelukast or montelukast alone. Any patients who have major contra-indications to steroids will be put into a separate observational group and receive montelukast only.

Drug regimens are prednisolone starting at 40 mg od nd tapered over 12 weeks. Montelukast 10mg od for 16 weeks.

The patients will be monitored weekly for 8 weeks then monthly for 4 months.

At least 20 patients will be enrolled in each group.

The patients will be closely observed for adverse effects, and any who deteriorate will receieve additional steroid according to the protocol. Any who develop new nerve function impairment will be removed from the trial and given a full course of prednisolone.

Analysis will be done on an intention to treat basis and will look for any statistically significant difference in ENL score at 2 weeks, 12 weeks and 24 weeks, or a difference in the number of patients who develop new nerve function impairment, as well as the incidence and severity of any adverse effects in each group.

ELIGIBILITY:
Inclusion Criteria:

* MB leprosy
* ENL reaction
* age 15-65
* weight >35kg
* patient willing to participate,including agrees to investigations and admission
* adequate past records
* no steroid received in past 4 weeks

Exclusion Criteria:

* pregnant or breast feeding
* other active serious infection
* history of intolerance to concerned drug
* known or suspected immunodeficiency
* needs high dose steroid for other condition
* recent new nerve funcion impairment
* recent hepatitis or impaired liver function
* thrombocytopenia, moderate or severe renal impairment
* received high dose clofazimine in past 3 months

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2006-12; Study Completion 2009-06

PRIMARY OUTCOMES:
decrease in ENL score
absence of new nerve function impairment
incidence of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Abdul H Salim, MBBS, Principal Investigator — Damien Foundation Bangladesh
Locations (1):
- Danish Bangladesh Leprosy Mission Hospital, Nilphamari, Nilphamari, Bangladesh